CLINICAL TRIAL: NCT05833906
Title: A Randomized, Single-blind, Placebo-controlled, Single/Multiple Dose, Dose Escalation, Phase 1 Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetic Characteristics of CKR-051 After Transdermal Administration in Healthy Male Subjects.
Brief Title: Safety, Tolerability, and Pharmacokinetic Evaluations of CKR-051 After Transdermal Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CK Regeon Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: COSMOS-21-RegenT-1
Record Dates: First submitted 2023-03-23; First posted 2023-04-27 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKR-051 SAD (Experimental): Participants will be administrated a single dermal dose of CKR-051 at various ascending dose levels or matching placebo for 1 day.
  Interventions: Drug: CKR-051 Dose 1; Drug: CKR-051 Dose 2; Drug: CKR-051 Dose 3; Drug: CKR-051 Dose 4; Drug: Placebo
- CKR-051 MAD (Experimental): Participants will be administrated a single dermal dose of CKR-051 at various ascending dose levels or matching placebo for 21 day.
  Interventions: Drug: CKR-051 Dose 2; Drug: CKR-051 Dose 3; Drug: CKR-051 Dose 4; Drug: Placebo

INTERVENTIONS:
Drug: CKR-051 Dose 1 — Subjects will be administered 5 g of CKR-051.
  Arms: CKR-051 SAD
Drug: CKR-051 Dose 2 — Subjects will be administered 10 g of CKR-051.
Drug: CKR-051 Dose 3 — Subjects will be administered 10 g of CKR-051.
Drug: CKR-051 Dose 4 — Subjects will be administered 10 g of CKR-051.
Drug: Placebo — Placebo comparator.

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of CKR-051 in healthy participants.

This study aiming to develop an agent for skin regeneration; potential treatments include acute and chronic wounds (c.f. Diabetic foot ulcers).

ELIGIBILITY:
Key Inclusion Criteria:

* Age 19 years to 60 years (Healthy male)
* Body weight 55 kg to 90 kg and BMI 19 kg/m^2 to 29 kg/m^2
* Do not have skin disease or skin damage (including scars or tattoos) or excessive body hair at the drug application site
* Must be suitable by a subject by medical evaluation including physical examination, laboratory tests, questionnaire, etc.

Key Exclusion Criteria:

* History of clinically significant hepatobiliary, kidney, nervous, immune, respiratory, digestive, endocrine, blood/tumor, cardiovascular, urinary, mental, dermatological diseases, etc.
* With tattoos, dermatitis, pigmentation, dermatitis, etc., or damaged skin at the site of clinical trial drug administration
* Drug hypersensitivity reactions and history (Aspirin, antibiotics, etc.)
* History of drug abuse and positive urine screening test
* eGFR (CKD-EPI) < 60 mL/min/1.73m^2
* AST/ALT > 1.5 UNL
* Alcohol > 21 units/week
* Smoker
* Eating food containing a grapefruit
* Caffeine > 5 units/day

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
SAD : Safety and tolerability (Numeric pain rating scale) | Day 1
  Score 0 to 7. Higher scores mean a worse outcome. 0 (No irritation); 1 (Minimal erythema); 2 (Erythema and papule); 3 (Palpable erythema and papule); 4 (Palpable edema); 5 (Edema, erythema and papule); 6 (Vesicular eruption); 7 (Spreading beyond the test area).
MAD : Safety and tolerability (Numeric pain rating scale) | Day 1 to Day 21 (Everyday)
  Score 0 to 7. Higher scores mean a worse outcome. 0 (No irritation); 1 (Minimal erythema); 2 (Erythema and papule); 3 (Palpable erythema and papule); 4 (Palpable edema); 5 (Edema, erythema and papule); 6 (Vesicular eruption); 7 (Spreading beyond the test area).

SECONDARY OUTCOMES:
SAD : Pharmacokinetics (Cmax) | Day 1
  Assessment of the peak plasma concentration of CKR-051
SAD : Pharmacokinetics (AUC) | Day 1
  Assessment of the plasma area under the curve of CKR-051
SAD : Pharmacokinetics (Tmax) | Day 1
  Assessment of the time to Cmax of CKR-051
SAD : Pharmacokinetics (t1/2) | Day 1
  Assessment of the total elimination half life of CKR-051
SAD : Pharmacokinetics (Vz/F) | Day 1
  Assessment of the volume of distribution of CKR-051
SAD : Pharmacokinetics (CL/F) | Day 1
  Assessment of the clearance of CKR-051
MAD : Pharmacokinetics (Cmax) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the peak plasma concentration of CKR-051
MAD : Pharmacokinetics (AUC) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the plasma area under the curve of CKR-051
MAD : Pharmacokinetics (Tmax) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the time to Cmax of CKR-051
MAD : Pharmacokinetics (t1/2) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the total elimination half life of CKR-051
MAD : Pharmacokinetics (Vz/F) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the volume of distribution of CKR-051
MAD : Pharmacokinetics (CL/F) | Day 1, 7, 14, 18, 19, 20 and 21
  Assessment of the clearance of CKR-051

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea